CLINICAL TRIAL: NCT00199043
Title: Randomised Phase III Trial of Effectivity and Safety of Rasburicase Compared With Allopurinol for Treatment of Hyperuricemia in Patients With Acute Lymphoblastic Leukemia or High-Grade NHL With High Risk of Tumorlysis Syndrome (> 15 Yrs)
Brief Title: Treatment of Hyperuricemia With Rasburicase in Patients With Acute Lymphoblastic Leukemia or High Grade Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Study Coordinator, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL08
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Adult Acute Lymphocytic Leukemia; High-grade Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin | interventions — Allopurinol; rasburicase

ARMS (1):
- Only 1 arm (Experimental)
  Interventions: Drug: Allopurinol; Drug: Rasburicase

INTERVENTIONS:
Drug: Allopurinol
Drug: Rasburicase

SUMMARY:
In this study the efficacy and tolerability of two approaches to treat and prevent hyperuricemia is tested in patients with acute lymphoblastic leukemia or high-grade lymphoma with high risk of tumor lysis syndrome. Both arms are compared by randomisation. In one arm patients receive during pre-phase chemotherapy conventional prophylaxis with allopurinol whereas in the other arm Rasburicase is used.

ELIGIBILITY:
Inclusion Criteria:

* patients of the GMALL B-ALL/NHL-Study 2002
* patients of the GMALL-Study 07/2003
* patients of the GMALL-Study Elderly 1/2003 which fulfill the following criteria:
* bulky disease (> 7.5 cm)
* high LDH (> 2 x UNL)
* uric acid >8 mg/dl/ >475µmol/L at diagnosis
* leukocytes > 30 000/µl

Exclusion Criteria:

* exclusion Criteria of the GMALL B-ALL/NHL Study 2002 or the GMALL-Study 07/2003 or GMALL-Elderly 1/2003 and:
* asthma or severe, live-threatening atopic allergy in history
* hypersensitivity against Uric acid
* Glucose-6-Phosphate-Dehydrogenase deficiency
* pretreatment with Rasburicase or Urikozyme™

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
renal function, uric acid, electrolytes, adverse events and mortality in pre-phase and the two following cycles of chemotherapy, time and dose compliance of chemotherapy | 3 weeks
  after cycle 1

SECONDARY OUTCOMES:
response rate, incidence of tumor lysis syndrome | 3 weeks
  after cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD,PhD, Study Chair — University Hospital of Frankfurt, Medical Dept. II
Locations (1):
- University Hospital, Medical Dept. II, Frankfurt, Germany